CLINICAL TRIAL: NCT04329923
Title: The PATCH Trial (Prevention And Treatment of COVID-19 With Hydroxychloroquine)
Acronym: PATCH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Cohort 1: slow accrual Cohort 2: Other studies showed no benefit Cohort 3: Study met pre-specificied futility analysis at planned second interim analysis
Sponsor: Ravi Amaravadi, MD (Other)
Responsible Party: Sponsor-Investigator, Ravi Amaravadi, MD, Associate Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 842838
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: There are 3 cohorts. All partcipants in of each the cohorts are randomized to one of two arms
Who Masked: Participant, Care Provider, Investigator
Masking Description: Cohorts 1 and 3 are double-blind placebo control cohorts. Cohort 2 is an open label randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 HCQ (Active Comparator): COVID-19 PCR+ patients quarantined at home randomized to this arm will be treated with hydroxychloroquine 400 mg twice a day for up to 14 days
  Interventions: Drug: Hydroxychloroquine Sulfate 400 mg twice a day
- Cohort 1 Placebo (Placebo Comparator): COVID-19 PCR+ patients quarantined at home randomized to this arm will be treated with placebo twice a day for up to 14 days. Crossover is allowed if symptoms worsen after 7 days of treatment.
  Interventions: Drug: Placebo oral tablet
- Cohort 2 HCQ high dose (Experimental): Hospitalized COVID-19 PCR+ patients randomized to this arm will be treated with hydroxychloroquine 600 mg twice a day for up to 14 days
  Interventions: Drug: Hydroxychloroquine Sulfate 600 mg twice a day
- Cohort 2 HCQ low dose (Active Comparator): Hospitalized COVID-19 PCR+ patients randomized to this arm will be treated with hydroxychloroquine 600 mg once a day for up to 7 days
  Interventions: Drug: Hydroxychloroquine Sulfate 600 mg once a day
- Cohort 3 HCQ (Experimental): Health care workers at high risk of contracting COVID-19 randomized to this arm will be treated with hydroxychloroquine 600 mg once a day for 2 months
  Interventions: Drug: Hydroxychloroquine Sulfate 600 mg once a day
- Cohort 3 Placebo (Placebo Comparator): Health care workers at high risk of contracting COVID-19 randomized to this arm will be treated with placebo for 2 month. Crossover is allowed if subject becomes SARS-CoV2 positive.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 400 mg twice a day — Antimalarial compound
  Other Names: Plaquenil
  Arms: Cohort 1 HCQ
Drug: Hydroxychloroquine Sulfate 600 mg twice a day — Antimalarial compound
  Other Names: Plaquenil
  Arms: Cohort 2 HCQ high dose
Drug: Hydroxychloroquine Sulfate 600 mg once a day — Antimalarial compound
  Other Names: Plaquenil
  Arms: Cohort 2 HCQ low dose; Cohort 3 HCQ
Drug: Placebo oral tablet — Placebo
  Other Names: Placebo
  Arms: Cohort 1 Placebo; Cohort 3 Placebo

SUMMARY:
The PATCH trial (Prevention And Treatment of COVID-19 with Hydroxychloroquine) is funded investigator-initiated trial that includes 3 cohorts. Cohort 1: a double-blind placebo controlled trial of high dose HCQ as a treatment for home bound COVID-19 positive patients; Cohort 2: a randomized study testing different doses of HCQ in hospitalized patients; Cohort 3: a double blind placebo controlled trial of low dose HCQ as a preventative medicine in health care workers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old (Sub-studies 2 and 3)
* Competent and capable to provide informed consent
* Have access to a smart device such as a cell phone, tablet, laptop computer with necessary data/internet accessibility
* Subjects meeting the following criteria by Sub-Study

Sub-Study 1:

* Age ≥40 years since the risk of prolonged disease that progresses to severe COVID-19 disease increases with age.
* PCR-positive for the SARS-CoV2 virus
* (Fever, and cough, or Fever and shortness of breath,
* ≤4 days since the first symptoms of COVID-19 and date of testing
* Not taking azithromycin
* Not requiring hospitalization and is sent home for quarantine.
* Must live within 30 miles of HUP or Penn Presbytarian Medical Center to facilitate drop-off of medication
* Must own a working computer, or smartphone and have internet access
* Must be willing to fill out a daily symptom diary
* Must be available for a daily phone call,
* Must take their own temperature twice a day
* Must be willing to report the observed symptoms and development of COVID-19 in the co-inhabitants of the residence at which the quarantine will be served.

Sub-Study 2 Hospitalized non-ICU service patients.

* PCR-positive for SARS-CoV-2
* Patients admitted to a floor bed at Hospital of the University of Pennsylvania or Penn Presbyterian.
* One or more of the following risk factors for progression to severe disease including: immunocompromising conditions, structural lung disease, hypertension, coronary artery disease, diabetes, age > 60, ferritin > 850, CRP > 6, D-dimer > 1000 Sub-Study 3 Health Care Worker Prevention
* Emergency Medicine or Infectious Disease Team physician or nurse at HUP or PPMC
* ≥20 hours per week of clinical work scheduled in the coming 2 months during the COVID-19 pandemic
* No fever, cough, or shortness of breath in the past 2 weeks
* Willing to report compliance with HCQ in the form of a diary
* Patients must be able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.

Exclusion Criteria <18 years of age

* Prisoners or other detained persons
* Allergy to hydroxychloroquine Pregnant or lactating or positive pregnancy test
* Receiving any treatment drug for 2019-ncov within 14 days prior to screening evaluation (off label, compassionate use or trial related).
* Co-enrollment onto another COVID-19 study is not allowed unless there is approval by the Medical Monitor in consultation with the PI and EM and ID sub-I leaders.
* Known history of retinal disease including but not limited to age related macular degeneration.
* Taking any of the following medications that prolong Qtc:

Chlorpromazine.Haloperidol, Droperidol, Quetiapine, Olanzapine. Amisulpride. Thioridazine

* History of interstitial lung disease or chronic pneumonitis unrelated COVID-19.
* Due to risk of disease exacerbation patients with porphyria or psoriasis are ineligible unless the disease is well controlled and they are under the care of a specialist for the disorder who agrees to monitor the patient for exacerbations.
* Patients with serious intercurrent illness that requires active infusional therapy, intense monitoring, or frequent dose adjustments for medication including but not limited to infectious disease, cancer, autoimmune disease, cardiovascular disease.
* Patients who have undergone major abdominal, thoracic, spine or CNS surgery in the last 2 months, or plan to undergo surgery during study participation.
* Patients receiving cytochrome P450 enzyme-inducing anticonvulsant drugs (i.e. phenytoin, carbamazepine, Phenobarbital, primidone or oxcarbazepine) within 4 weeks of the start of the study treatment
* History or evidence of increased cardiovascular risk including any of the following:
* Left ventricular ejection fraction (LVEF) < institutional lower limit of normal. Baseline echocardiogram is not required.
* A QT interval corrected for heart rate using the Frederica formula > 500 msec (Sub-study 2)
* Current clinically significant uncontrolled arrhythmias. Exception: Subjects with controlled atrial fibrillation
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to enrollment
* Current ≥ Class II congestive heart failure as defined by New York Heart Association

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will publish our results in a peer-reviewed journal and make available de-identified data for additional analysis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after study completion
Access Criteria: Open access

REFERENCES:
- [Result] Abella BS, Jolkovsky EL, Biney BT, Uspal JE, Hyman MC, Frank I, Hensley SE, Gill S, Vogl DT, Maillard I, Babushok DV, Huang AC, Nasta SD, Walsh JC, Wiletyo EP, Gimotty PA, Milone MC, Amaravadi RK; Prevention and Treatment of COVID-19 With Hydroxychloroquine (PATCH) Investigators. Efficacy and Safety of Hydroxychloroquine vs Placebo for Pre-exposure SARS-CoV-2 Prophylaxis Among Health Care Workers: A Randomized Clinical Trial. JAMA Intern Med. 2021 Feb 1;181(2):195-202. doi: 10.1001/jamainternmed.2020.6319. PMID 33001138

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 HCQ | Cohort 1 Placebo | Cohort 2 HCQ High Dose | Cohort 2 HCQ Low Dose | Cohort 3 HCQ | Cohort 3 Placebo
Started | 17 | 17 | 4 | 3 | 66 | 66
Completed | 16 | 13 | 3 | 2 | 64 | 61
Not Completed | 1 | 4 | 1 | 1 | 2 | 5
Not completed — Withdrawal by Subject | 1 | 4 | 1 | 1 | 1 | 1
Not completed — early termination of study | 0 | 0 | 0 | 0 | 1 | 2
Not completed — positive SARS-COV2 PCR at baseline | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 HCQ | Cohort 1 Placebo | Cohort 2 HCQ High Dose | Cohort 2 HCQ Low Dose | Cohort 3 HCQ | Cohort 3 Placebo | Total
Number analyzed (Participants) | 17 | 17 | 4 | 3 | 66 | 66 | 173
Age, Continuous [Median (Full Range); unit: years] | 56 [43 to 77] | 49 [40 to 80] | 65 [41 to 79] | 48 [30 to 55] | 31 [20 to 66] | 34 [23 to 62] | 40 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 2 | 3 | 54 | 33 | 113
  Male | 5 | 8 | 2 | 0 | 12 | 33 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 11 | 3 | 3 | 3 | 1 | 29
  White | 6 | 3 | 1 | 0 | 55 | 56 | 121
  More than one race | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Unknown or Not Reported | 3 | 3 | 0 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Release From Quarantine Time
Description: Cohort 1 (home quarantined COVID-19 patients): Median time to release from quarantine by meeting the following criteria: 1) No fever for 72 hours 2) improvement in other symptoms and 3) 7 or 10 days (depending on CDC guidance at the time) have elapsed since the beginning of symptom onset.
Time Frame: until quarantine release or hospitalization
Population: randomized patients that were released from quarantine on study
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 1 HCQ | Cohort 1 Placebo
Number analyzed (Participants) | 15 | 13
days | 8 [4 to 19] | 11 [4 to 18]
Statistical Analysis 1: Comparison: Cohort 1 HCQ vs Cohort 1 Placebo; Test type: Superiority; p = 0.28, Regression, Cox; Cox Proportional Hazard = 0.58

2. Primary Outcome: Time to Hospital Discharge
Description: Cohort 2 (hospitalized COVID-19 patients): median number of days until hospital discharge
Time Frame: until hospital discharge
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 2 HCQ High Dose | Cohort 2 HCQ Low Dose
Number analyzed (Participants) | 4 | 3
days | 5.5 [2 to 15] | 4 [3 to 15]

3. Primary Outcome: Number of Health Care Workers Who Developed SARS-COV-2 Infection
Description: Cohort 3 Physicians and nurse prophylaxis: Rate of COVID-19 infection at 2 months
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3 HCQ | Cohort 3 Placebo
Number analyzed (Participants) | 64 | 61
Participants | 4 | 4

4. Secondary Outcome: Rate of Housemate Infection
Description: Cohort 1 rate of participant-reported secondary infection of housemates
Time Frame: until quarantine release, or approximately <20 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 HCQ | Cohort 1 Placebo
Number analyzed (Participants) | 17 | 17
Participants | 2 | 2

5. Secondary Outcome: Rate of Hospitalization
Description: Cohort 1 rate of hospitalization
Time Frame: until quarantine release
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 HCQ | Cohort 1 Placebo
Number analyzed (Participants) | 17 | 17
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: All adverse events were grade 1-2 by CTCAE v5.0
Arm/Group | Cohort 1 HCQ | Cohort 1 Placebo | Cohort 2 HCQ High Dose | Cohort 2 HCQ Low Dose | Cohort 3 HCQ | Cohort 3 Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/4 | 0/3 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/17 | 0/4 | 0/3 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 6/17 | 3/17 | 0/4 | 1/3 | 29/66 | 15/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 HCQ (N=17) | Cohort 1 Placebo (N=17) | Cohort 2 HCQ High Dose (N=4) | Cohort 2 HCQ Low Dose (N=3) | Cohort 3 HCQ (N=66) | Cohort 3 Placebo (N=66)
hospitalization (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The patient developed progressive symptoms of COVID-19 and was hospitalized briefly for supplemental oxygen
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 HCQ (N=17) | Cohort 1 Placebo (N=17) | Cohort 2 HCQ High Dose (N=4) | Cohort 2 HCQ Low Dose (N=3) | Cohort 3 HCQ (N=66) | Cohort 3 Placebo (N=66)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Anorexia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 21 (21) | 8 (8)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 5 (5)

LIMITATIONS AND CAVEATS:
Sub-study 1 was terminated early after the first interim analysis due to slow accrual Sub-study 2 was terminated early after the first 7 patients based on the recommendation of UPenn research oversight committees Sub-study 3 was terminated early due to meeting futility criteria on a pre-specified second interim analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT04329923/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT04329923/SAP_002.pdf